CLINICAL TRIAL: NCT06856798
Title: Construction of a Efficacy Stratification Prognostic and Prediction Model for Perioperative Immunotherapy in Non - Small Cell Lung Cancer Based on Multi - Omics Biomarkers
Brief Title: Construction of a Prognostic and Prediction Model for Perioperative Immunotherapy in NSCLC: a Multi - Omics Perspective
Status: Not yet recruiting | Type: Observational
Sponsor: Ziming Li (Other)
Responsible Party: Sponsor-Investigator, Ziming Li, Chief of the Oncology Department, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Other Study IDs: IS25015
Record Dates: First submitted 2025-02-10; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: NSCLC Stage IIIA/B; NSCLC Stage II
Keywords: Multi - Omics Biomarkers; Immunotherapy; Perioperative; ctDNA; MRD
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Boold，tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PD-1/PD-L1 neoadjuvant therapy group: Patients with non - small cell lung cancer who are negative for driver genes such as EGFR and ALK and receive neoadjuvant immunotherapy

SUMMARY:
This research focuses on exploring biomarkers for the application of PD - 1/PD - L1 immune checkpoint inhibitors in the perioperative immunotherapy of lung cancer. Multi - index tests are conducted on tissues prior to treatment, as well as blood samples at baseline and during the treatment course. The goal is to identify biomarkers capable of predicting the efficacy of neoadjuvant and adjuvant immunotherapies. Additionally, by integrating these multiple - index data into models, patients are to be stratified based on their potential benefits from perioperative immunotherapy, providing personalized guidance for clinical decision - making.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC, clinical tumor stage II-IIIB
* Without EGFR/ALK gene mutation
* Patient 18 years or older.
* Scheduled for neoadjuvant immunotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-1
* Life expectancy ≥ 12 weeks.
* Patient able to understand and sign written informed consent.

Exclusion Criteria:

* With other cancers (excluding NSCLC or skin cancer other than melanoma, or cancers treated curatively with follow up of more than 5 years without recurrence).
* With history of chemotherapy or radiotherapy (including pre - operative and post - operative adjuvant chemotherapy and radiotherapy) or systemic anti - tumor treatment.
* with autoimmune diseases unsuitable for PD - 1 monoclonal antibody treatment, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain - Barré syndrome, or multiple sclerosis.
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude), inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non - small cell lung cancer who are negative for driver genes such as EGFR and ALK and receive neoadjuvant immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-03-09 (Estimated); Study Completion 2028-02-09 (Estimated)

PRIMARY OUTCOMES:
Pathological response after immune neoadjuvant therapy | From enrollment to surgery at 18 weeks
  The primary evaluation indicators are pathological complete response (pCR) and major pathological response (MPR). MPR refers to the residual tumor cells in the surgically resected specimens being ≤ 10%, while pCR requires the complete disappearance of tumor cells.

SECONDARY OUTCOMES:
2-year Progression-Free Survival(PFS1) | PFS of patients from the time of enrollment until two years
  Mainly evaluate the PFS of patients from the time of enrollment until two years later.
2-year Progression-Free Survival(PFS2) | PFS from the start of adjuvant immunotherapy to 2 years.
  Mainly evaluate the patient's PFS from the start of adjuvant immunotherapy to 2 years.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu J, Wan R, Cai Y, Cai S, Wu L, Li B, Duan J, Cheng Y, Li X, Wang X, Han L, Wu X, Fan Y, Yu Y, Lv D, Shi J, Huang J, Zhou S, Han B, Sun G, Guo Q, Ji Y, Zhu X, Hu S, Zhang W, Wang Q, Jia Y, Wang Z, Song Y, Wu J, Shi M, Li X, Han Z, Liu Y, Yu Z, Liu AW, Wang X, Zhou C, Zhong D, Miao L, Zhang Z, Zhao H, Yang J, Wang D, Wang Y, Li Q, Zhang X, Ji M, Yang Z, Cui J, Gao B, Wang B, Liu H, Nie L, He M, Jin S, Gu W, Shu Y, Zhou T, Feng J, Yang X, Huang C, Zhu B, Yao Y, Yu J, Yao S, Shen R, Wang Z, Wang J. Circulating tumor DNA-based stratification strategy for chemotherapy plus PD-1 inhibitor in advanced non-small-cell lung cancer. Cancer Cell. 2024 Sep 9;42(9):1598-1613.e4. doi: 10.1016/j.ccell.2024.08.013. PMID 39255777
- [Background] Ai X, Jia B, He Z, Zhang J, Zhuo M, Zhao J, Wang Z, Zhang J, Fan Z, Zhang X, Li C, Jin F, Li Z, Ma X, Tang H, Yan X, Li W, Xiong Y, Yin H, Chen R, Lu S. Noninvasive early identification of durable clinical benefit from immune checkpoint inhibition: a prospective multicenter study (NCT04566432). Signal Transduct Target Ther. 2024 Dec 16;9(1):350. doi: 10.1038/s41392-024-02060-3. PMID 39676097